CLINICAL TRIAL: NCT06324474
Title: Clinical and Immunological Evaluation of Hyaluronic Acid Topical Application in Non-surgical Treatment of Periodontitis
Brief Title: Clinical and Immunological Evaluation of HA in Treatment of Periodontitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sana'a University (Other)
Responsible Party: Principal Investigator, ghada almuqayad, Principal Investigator,, Sana'a University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HA treatment of periodontitis
Record Dates: First submitted 2023-11-25; First posted 2024-03-22 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Hyaluronic Acid; Tooth Exfoliation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- scaling and root planning with Hyaluronic acid application (Experimental): patients will receive Hyaluronic acid topical gel after scaling and root planning at first week and receive the gel after one week
  Interventions: Drug: Hyaluronic acid; Behavioral: scaling and root planning
- scaling and root planning only (Experimental): patients will receive scaling and root planning only
  Interventions: Behavioral: scaling and root planning

INTERVENTIONS:
Drug: Hyaluronic acid — Gengigel syringe containing 1ml of 0.8% HA
  Other Names: HA syringe
  Arms: scaling and root planning with Hyaluronic acid application
Behavioral: scaling and root planning — scaling and root planning using ultrasonic scaler

SUMMARY:
To evaluate the immunological effectiveness of Hyaluronic acid as adjunction treatment to scaling and root planning and scaling and root planning alone.

Comparison between clinical measurement before and after treatment. Evaluate the level of IGF-1 in treated site as immunological marker if periodontal regeneration.

DETAILED DESCRIPTION:
Periodontal tissue represents a unique system, where the epithelial, non- mineralized, and mineralized connective tissues exist in harmony. This integrity is essential in providing an effective barrier against microbial invasion and preventing the destruction of underlying periodontal tissues by bacterial toxins and enzymes. However; it may lose during chronic inflammation associated with periodontal disease leading to detrimental effects upon the extracellular matrix components of underlying periodontal tissues, including collagens, proteoglycans, and glycosaminoglycans.

Periodontitis is a chronic multifactorial inflammatory disease associated with plaque biofilms and characterized by progressive destruction of the tooth- supporting apparatus. It is considered as an inflammatory condition of the periodontium, which includes an immune response and results in loss of supporting tissues of the teeth. It may affect the general health; a combination of mechanical and chemical treatment provides a good recovery. The etiology for this disease is the accumulation of bacterial plaque on the tooth surface that leads to marginal tissue inflammation, known as gingivitis which is reversable condition that may develop to periodontitis if not treated. ( A new periodontitis scheme has been adopted in which forms of disease previously recognized as 'chronic' or 'aggressive' are now grouped under a single category 'periodontitis' and are further characterized based on a multi-dimensional staging and grading system. Staging is largely dependent upon the severity of disease at presentation as well as on the complexity of disease management, while grading provides supplemental information about biological feature of the disease.

However, the final success rate of the treatment depends on the status and maintenance of oral hygiene. Signs and symptoms of periodontitis may include redness, swelling bleeding of gum, loss of attachment, halitosis and persistent metallic taste in the mouth.

Antibiotics are mandatory in some cases, systemic antibiotics somewhat are effective, no single antibiotic at concentrations achieved in body fluids inhibits all putative periodontal pathogens, indeed a combination of antibiotics may be necessary to eliminate all putative pathogen from some periodontal pockets. ( Topical application has the advantage that antibiotic agents are directed to their specific target areas; reduced drug dosage, increased drug concentration, and reduced side effects can be benefits of topical application. Unfortunately, some antibiotics when used topically induce superinfection and hypersensitivity reaction.

Hyaluronic acid (HA) is an indispensable component of intact, healthy gingiva, and oral mucosal tissue. It has many properties that make it ideal molecule for assisting wound healing by inducing early granulation tissue formation, inhibiting inflammation, promoting epithelial turnover, and also connective tissue angiogenesis. It has many important physiological and biological functions and plays a vital role in the functioning of extracellular matrix including those of periodontium.

Its application as adjunct to non-surgical periodontal treatment seems to have a beneficial effect on surrogate outcome variables of periodontal inflammation, thus; its emerging as a boon prospect in treatment of periodontitis.

Jain Y. proved on a research done on 2013 that 0.2% HA was effective agent on plaque induced gingivitis as an adjunct to scaling as compared to scaling alone, however; a study was done in 2015 in sub-gingival placement of 0.2 ml of 0.8% of HA along with scaling and root planning (SRP) had a significant improvement in both clinical and microbiological parameters when compared with the control site.

Gingival cervical fluid (GCF) is a physiological fluid as well as an inflammatory exudate originating from the gingival plexus of blood vessels in the gingival corium, subjacent to the epithelium lining of the dento-gingival space, Collection of GCF is non-invasive there for this approach has been extensively explored in the search for potential diagnostic biomarker of periodontal disease. Numerous cytokines are released from cells of the sulcular and junctional epithelium. Growth factors are biologically active polypeptides affecting the proliferation, chemotaxis, and differentiation of cells from epithelium, bone and connective tissue. They express their action by binding to specific cell surface receptors present on various target cells including osteoblast, cementoblast, and periodontal ligament fibroblast.

Insulin like growth factor (IGF-1) is a potent mitogenic protein which can enhance the osteogenic differentiation of periodontal ligament fibroblast.

The more the concentration of IGF-1 the more the cell proliferation as proven in a study of insulin like growth factor-1 promotes proliferation, migration and osteoblast differentiation of periodontal ligament stem cell.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy.
* at least 20 teeth and suffers from moderate <7mm to severe. >8mm.periodontitis with probing depth >5m and in the contralateral side.
* ability to attend to the clinic in a regular manner.

Exclusion Criteria:

* allergy to HA.
* Chronic disease.
* orthodontic treatment.
* Qat chewer and smokers.
* antibiotic in previous 3 months.
* supplements and mouthwash.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12-12 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Plaque Index | From Baseline to 12th weeks post intervention '' changes from baseline to 12th week"
  ranges from 0 to 3 score, where increasing in number indicates the worst case.
Changes in Gingival Index | From Baseline to 12th weeks post intervention '' changes from baseline to 12th week"
  Ranges from 0 to 3 stages, where increasing in number indicates the worst case.
Changes in Papillary Bleeding Index. | From Baseline to 12th weeks post intervention '' changes from baseline to 12th week"
  Ranges from 0 to 4 score, where increasing in number indicates the worst case
Periodontal Probing Depth | From Baseline to 12th weeks post intervention '' changes from baseline to 12th week"
  distance from the gingival margin to the base of the pocket
Clinical attachment loss | From baseline to 12th weeks post intervention "changes from baseline to 12th week
  Distance from cemento-enamel junction to the base of pocket
Changes in IGF-1 | From baseline to 12th weeks post intervention "changes from baseline to 12th week
  Through gingival cervical fluid serum collection

CONTACTS AND LOCATIONS:
Overall Officials: Ghada Almuqayad, BDS, Principal Investigator — Sana'a University
Locations (1):
- Sana'a university, Sanaa, Yemen

REFERENCES:
- [Background] Polepalle T, Srinivas M, Swamy N, Aluru S, Chakrapani S, Chowdary BA. Local delivery of hyaluronan 0.8% as an adjunct to scaling and root planing in the treatment of chronic periodontitis: A clinical and microbiological study. J Indian Soc Periodontol. 2015 Jan-Feb;19(1):37-42. doi: 10.4103/0972-124X.145807. PMID 25810591
- [Background] Al-Shammari NM, Shafshak SM, Ali MS. Effect of 0.8% Hyaluronic Acid in Conventional Treatment of Moderate to Severe Chronic Periodontitis. J Contemp Dent Pract. 2018 May 1;19(5):527-534. PMID 29807962
- [Background] Barros SP, Williams R, Offenbacher S, Morelli T. Gingival crevicular fluid as a source of biomarkers for periodontitis. Periodontol 2000. 2016 Feb;70(1):53-64. doi: 10.1111/prd.12107. PMID 26662482
- [Background] Alsakhawy SA, Baghdadi HH, El-Shenawy MA, Sabra SA, El-Hosseiny LS. Encapsulation of thymus vulgaris essential oil in caseinate/gelatin nanocomposite hydrogel: In vitro antibacterial activity and in vivo wound healing potential. Int J Pharm. 2022 Nov 25;628:122280. doi: 10.1016/j.ijpharm.2022.122280. Epub 2022 Oct 13. PMID 36243326
- [Background] Caton JG, Armitage G, Berglundh T, Chapple ILC, Jepsen S, Kornman KS, Mealey BL, Papapanou PN, Sanz M, Tonetti MS. A new classification scheme for periodontal and peri-implant diseases and conditions - Introduction and key changes from the 1999 classification. J Clin Periodontol. 2018 Jun;45 Suppl 20:S1-S8. doi: 10.1111/jcpe.12935. PMID 29926489
- [Background] Gontiya G, Galgali SR. Effect of hyaluronan on periodontitis: A clinical and histological study. J Indian Soc Periodontol. 2012 Apr;16(2):184-92. doi: 10.4103/0972-124X.99260. PMID 23055583
- [Background] Sahayata VN, Bhavsar NV, Brahmbhatt NA. An evaluation of 0.2% hyaluronic acid gel (Gengigel (R)) in the treatment of gingivitis: a clinical & microbiological study. Oral Health Dent Manag. 2014 Sep;13(3):779-85. PMID 25284557
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] Loe H. The Gingival Index, the Plaque Index and the Retention Index Systems. J Periodontol. 1967 Nov-Dec;38(6):Suppl:610-6. doi: 10.1902/jop.1967.38.6.610. No abstract available. PMID 5237684
- [Background] Dereka XE, Markopoulou CE, Vrotsos IA. Role of growth factors on periodontal repair. Growth Factors. 2006 Dec;24(4):260-7. doi: 10.1080/08977190601060990. PMID 17381067
- [Background] Al-Khateeb R, Olszewska-Czyz I. Biological molecules in dental applications: hyaluronic acid as a companion biomaterial for diverse dental applications. Heliyon. 2020 Apr 6;6(4):e03722. doi: 10.1016/j.heliyon.2020.e03722. eCollection 2020 Apr. PMID 32280803
- [Background] Papapanou PN, Sanz M, Buduneli N, Dietrich T, Feres M, Fine DH, Flemmig TF, Garcia R, Giannobile WV, Graziani F, Greenwell H, Herrera D, Kao RT, Kebschull M, Kinane DF, Kirkwood KL, Kocher T, Kornman KS, Kumar PS, Loos BG, Machtei E, Meng H, Mombelli A, Needleman I, Offenbacher S, Seymour GJ, Teles R, Tonetti MS. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S173-S182. doi: 10.1002/JPER.17-0721. PMID 29926951
- [Background] Van der Weijden GAF, Dekkers GJ, Slot DE. Success of non-surgical periodontal therapy in adult periodontitis patients: A retrospective analysis. Int J Dent Hyg. 2019 Nov;17(4):309-317. doi: 10.1111/idh.12399. Epub 2019 May 16. PMID 30942938
- [Background] Pradeep AR, Kumari M, Rao NS, Naik SB. 1% alendronate gel as local drug delivery in the treatment of Class II furcation defects: a randomized controlled clinical trial. J Periodontol. 2013 Mar;84(3):307-15. doi: 10.1902/jop.2012.110729. Epub 2012 May 3. PMID 22554293
- [Background] Ma S, Liu G, Jin L, Pang X, Wang Y, Wang Z, Yu Y, Yu J. IGF-1/IGF-1R/hsa-let-7c axis regulates the committed differentiation of stem cells from apical papilla. Sci Rep. 2016 Nov 11;6:36922. doi: 10.1038/srep36922. PMID 27833148
- [Background] Sukumar S, Drizhal I. Hyaluronic acid and periodontitis. Acta Medica (Hradec Kralove). 2007;50(4):225-8. PMID 18290544
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464